CLINICAL TRIAL: NCT02659644
Title: A Phase I Dose-Ranging Study of Oral L-citrulline in Steady-State Sickle Cell
Brief Title: A Study of Oral L-citrulline in Sickle Cell Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal Investigator moved to another institution
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Suvankar Majumdar, Associate Professor, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-0191
Record Dates: First submitted 2015-12-29; First posted 2016-01-20 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Citrulline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral citrulline (Experimental)
  Interventions: Drug: Oral L-citrulline

INTERVENTIONS:
Drug: Oral L-citrulline — There will be a total of 16 patients divided into 4 equal cohorts. The first 4 cohorts will be started on a 7 day oral regimen of twice daily L-citrulline. They will return to clinic on day #7 to evaluate nitric oxide metabolite levels and pharmacokinetic (PK) profile of citrulline. After PK analysis, the next cohort of patients will be given a higher or lower dose based on their weight and also based safety and tolerability. Of note, a PK analysis will be performed for each 4 patient cohort prior to starting citrulline for the subsequent cohort. Assessment for adverse events will be done at specified times throughout the study duration via both phone and clinic encounters.

SUMMARY:
Sickle cell disease is a genetic red blood cell disorder that can result in blocking of the small blood vessels from sickle shaped red blood cells. This causes pain, the main feature of sickle cell disease. Also, low amounts of nitric oxide can occur in sickle cell disease, a substance important for widening the blood vessel wall and therefore preventing blockage of the small blood vessels.

Citrulline is a drug that is known to increase nitric oxide. This is a phase I study of citrulline given by mouth to evaluate the safety, tolerability and appropriate dosing of this medication for individuals with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

1. Sickle cell disease genotypes (HbSS, HbS/β-thalassemia
2. HbS/β+thalassemia, HbSC)
3. Patients with sickle cell disease aged 10 to 25 years old
4. Patients ages 10 through 17 years of age, whose parents have signed permission, and who provide signed patient assent themselves
5. Patients 18 through 25 years of age who provide signed consent.

Exclusion Criteria:

1. Presence of any acute illness defined by fever >100.4°F within the past 48 hours
2. Presence of sickle cell pain crisis defined by the presence of pain requiring oral or parental opioid therapy.
3. Presence of acute chest syndrome or presence of any other complication related to sickle cell disease requiring hospitalization such as splenic sequestration, hepatic sequestration, stroke, avascular necrosis of the hip/shoulder, acute priapism, and patients with diabetes etc.
4. Severe anemia (hemoglobin < 5g/dL)
5. History of red blood cell transfusion within the last 14 days
6. Systemic steroid therapy within the last 48 hours
7. Pregnant (as confirmed by a negative urine pregnancy test) or lactating female
8. Alanine/aspartate transferase >2x upper limit of normal laboratory range for age.
9. Elevated serum creatinine: Age 6 to 13 years > 0.9 mg/dL, Age 14-17 years 1.0 mg/dL, Age >18 years >1.5mg/dL
10. Patients with an inability to give assent (ages 10 to 17 years) or consent (ages 18 through 25 years) will be excluded
11. History of diabetes due to risk of electrolyte imbalance

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Peak plasma citrulline concentration (Cmax) | 7 days
Rate of citrulline appearance (Rapp) | 7 days
Constant of citrulline removal (krem) | 7 days
Volume of distribution | 7 days
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 7 days

SECONDARY OUTCOMES:
Level of nitric oxide | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwedhelm E, Maas R, Freese R, Jung D, Lukacs Z, Jambrecina A, Spickler W, Schulze F, Boger RH. Pharmacokinetic and pharmacodynamic properties of oral L-citrulline and L-arginine: impact on nitric oxide metabolism. Br J Clin Pharmacol. 2008 Jan;65(1):51-9. doi: 10.1111/j.1365-2125.2007.02990.x. Epub 2007 Jul 27. PMID 17662090
- [Background] Moinard C, Nicolis I, Neveux N, Darquy S, Benazeth S, Cynober L. Dose-ranging effects of citrulline administration on plasma amino acids and hormonal patterns in healthy subjects: the Citrudose pharmacokinetic study. Br J Nutr. 2008 Apr;99(4):855-62. doi: 10.1017/S0007114507841110. Epub 2007 Oct 22. PMID 17953788